CLINICAL TRIAL: NCT04310410
Title: Feasibility of Combined Focused Ultrasound and Radiotherapy Treatment in Patients With Painful Bone Metastasis - the PRE-FURTHER Study -
Brief Title: Feasibility of Combined Focused Ultrasound and Radiotherapy Treatment in Patients With Painful Bone Metastasis
Acronym: PRE-FURTHER
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Isala (Other)
Responsible Party: Principal Investigator, Helena M Verkooijen, Principal Investigator, UMC Utrecht
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: NL68441.041.19
Record Dates: First submitted 2019-09-24; First posted 2020-03-17 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Bone Metastases; Bone Neoplasm; Bone Lesion; Bone Cancer; Pain; Cancer Induced Bone Pain; Radiation Toxicity; Quality of Life; Tumor; Neoplasm Metastasis
Keywords: Bone metastases; Cancer Induced Bone Pain; Pain palliation; Radiotherapy; Radiation oncology; MR-HIFU; MRI-guided high intensity focused ultrasound; Focused ultrasound; HIFU
MeSH Terms: conditions — Bone Neoplasms; Pain; Radiation Injuries; Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Prospective case series (n = 6 - 10), stage I and IIA study according to the Innovation, Development, Evaluation, Assessment and Long term evaluation (IDEAL) recommendations. The study will be performed in male and female adult (≥ 18 years) cancer patients capable of giving informed consent and referred for EBRT of painful bone metastases (Numerical Rating Scale (NRS) ≥ 4).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined Focused Ultrasound and Radiotherapy (Experimental): Combination of focused ultrasound and external beam radiotherapy
  Interventions: Combination Product: combined radiotherapy and MR-HIFU

INTERVENTIONS:
Combination Product: combined radiotherapy and MR-HIFU — Following standard EBRT (single or multiple fraction), patients will receive one MR-HIFU treatment with the Profound Sonalleve MR-HIFU device on the most painful of their bone metastases. This treatment will take place in a short time frame of 3 hours to maximum 4 days. Patients will be followed up until 4 weeks after treatment. During follow-up they will be phoned around day 3, 7, 14, 21 and 28 to retrieve pain scores, pain medication and (serious) adverse events. At day 3 the patient's experience with the combined treatment will also be inquired.

SUMMARY:
The PRE-FURTHER study aims to evaluate the feasibility of the combined treatment with radiotherapy and focussed ultrasound for pain palliation in patients with painful bone metastases, and to optimize the combined treatment logistics. Six to ten patients will be included according to in- and exclusion criteria.

DETAILED DESCRIPTION:
Rationale: Metastatic bone pain strongly interferes with quality of life and daily functioning of patients with advanced cancer. Pain palliation may be improved by including magnetic resonance image guided high intensity focused ultrasound (MR-HIFU) in addition to External Beam Radiotherapy (EBRT). For this purpose, feasibility and optimal logistics of the combined treatment need to be evaluated.

Objective: The PRE-FURTHER project aims to evaluate the feasibility of the combined EBRT and MR-HIFU treatment for relief of metastatic bone pain, and to optimize the combined treatment logistics.

Study design: The PRE-FURTHER study is a prospective case series, stage I and IIA study according to the Innovation, Development, Evaluation, Assessment and Long term evaluation (IDEAL) recommendations. 6-10 patients will receive MR-HIFU treatment following standard EBRT.

Endpoints: The main outcome of this study is the feasibility of the procedure, in terms of planability as well as patient-tolerability of the combined treatment within a short time frame (3 hours - 4 days interval). In addition, pain relief and safety of the combined procedure will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with age ≥ 18 years
* Patient capable of giving informed consent and able to attend study visits
* Uncomplicated painful bone metastases
* Weight <140kg and able to fit in the MRI gantry
* Radiologic evidence of bone metastases from any solid tumor
* Pain is localized to the targeted area, or is likely to be referred pain arising from the targeted area
* Pain related to the target lesion is refractory to less invasive treatments for pain relief
* Multiple metastatic lesions, with one predominantly painful lesion (>=2 points higher pain score than other lesions). The lesion should be clearly distinguishable from other painful lesions.
* Device accessible tumors: extremities (excluding joints), pelvis, shoulders, posterior vertebral spine below L5, in selected cases ribs and sternum
* Target lesion maximum dimension ≤ 8cm
* Intended target volume visible by non-contrast MR imaging
* Distance between target and skin ≥ 1cm
* Numeric Rating Scale (NRS) score >= 4 or equivalent
* Life expectancy >3 months

Exclusion Criteria:

* Planned treatment lesion is a primary bone tumor or due to lymphoma, multiple myeloma, or leukemia.
* Communication barrier present
* Patient enrolled in another clinical study related to bone metastases treatment or pain relief treatment
* Unable to tolerate required stationary position during treatment despite adequate pain medication
* Need for surgery
* Pregnant woman
* Pain related to target lesion is predominantly due to fracture or impending fracture
* Pain related to target lesion is due to involvement of a neighboring major nerve by the metastatic tumor (cord or nerve compression)
* Target < 3cm from bladder / bowel / nerve along the beam path and < 1cm in the plane orthogonal to the beam
* Target in contact with hollow viscera
* Target located in skull, joints, ribs (when HIFU beam overlapping with lung), spine (excluding sacrum which is allowed) or in most cases sternum
* Internal or external fixation device along the proposed HIFU beam path or at the target
* MRI contraindicated (e.g. paramagnetic implants, pacemaker, claustrophobia)
* MRI contrast agent contraindicated (e.g. previous anaphylaxis or Glomerular Filtration Rate < 20 ml/min/1.73m2)
* Sedation contraindicated
* Previous surgery or minimally invasive treatment at targeted site within the last three months
* Clinically relevant medical history or abnormal physical findings that could interfere with the safety of the participant as judged by the treating physician or investigator
* Karnofsky performance score (KPS) < 60%
* Oligometastatic disease planned for curative treatment
* Indication for stereotactic radiotherapy (e.g. patients with radioresistant histology such as renal cell, melanoma, sarcoma metastases)
* History of photodermatoses (of the skin overlying the target area)
* Need for remineralisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of combined treatment with EBRT and MR-HIFU - Patient tolerance: questionnaire | 4 weeks
  The main outcome of this study is the feasibility of the combined procedure in terms of patient tolerance and hospital logistics. Patient tolerance will be assessed using a Patient Reported Experience Measure questionnaire.
Feasibility of combined treatment with EBRT and MR-HIFU - hospital logistics | 4 weeks
  The main outcome of this study is the feasibility of the combined procedure in terms of patient tolerance and hospital logistics. Hospital logistics will be assessed by analysing comments of the treating physicians and research staff on the problems that occurred during treatment planning, and whether extra hospital visits that were needed.

SECONDARY OUTCOMES:
Patient reported pain scores. | at 3 days, and at 1, 2, 3 and 4 weeks
  Patient reported pain scores will be based on a Numeric Rating Scale (from 0 to 10 with 0 being no pain and 10 being the worst pain imaginable) from the Brief Pain Inventory (BPI) questionnaire [Cleeland 1994].
(Serious) adverse events | at 3 days, and at 1, 2, 3 and 4 weeks
  Toxicity/safety of the combined treatment will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Helena M Verkooijen, MD, PhD, Principal Investigator — UMC Utrecht
Locations (2):
- Netherlands (2):
  - Isala Klinieken Zwolle, Zwolle, Overijsel
  - University Medical Center Utrecht, Utrecht

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT04310410/Prot_SAP_000.pdf